CLINICAL TRIAL: NCT07073118
Title: Safety and EffecTiveness of the Silk Vista Flow DiverteR in the TrEatment of Unruptured IntracrAnial AneurysMs
Acronym: STREAM
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Balt Extrusion (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2025/023
Record Dates: First submitted 2025-07-08; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Ruptured and Unruptured Intracranial Aneurysms
Keywords: Intracranial aneurism; flow-diverter stent
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with unruptured intracranial aneurysm: Patients aged ≥ 18 and ≤ 80 years old, with at least one unruptured intracranial aneurysm intended to be treated with Silk Vista
  Interventions: Device: Endovascular treatment with placement of a flow-diverting stent

INTERVENTIONS:
Device: Endovascular treatment with placement of a flow-diverting stent — Flow diverter stents (FDS) are braided stents with specific porosity that promotes the flow redirection within the parent vessel and outside the aneurysm sac, and the endothelialization. The FDS placed in the parent artery and covering the aneurysm sac will promote the intra-aneurysmal blood stagnation and parent vessel wall healing. All of these promoting, the aneurysm's thrombosis and ist regression

SUMMARY:
Intracranial aneurysms (IA) are abnormal outpouchings of cerebral arteries' walls that occur mostly in arteries found in the Circle of Willis and the middle cerebral artery bifurcation with a risk of rupture leading to subarachnoid hemorrhage (SAH) and potentially death. If IA is treated before rupture, survival rates improve dramatically. The IA can be treated with endovascular technique (coiling or stenting). Specifically, the parent artery reconstruction with a flow-diverter stent allows the treatment of a wide range of aneuryms with high rate of aneurysm occlusion. However, during follow-up, up to 15% of FD present deformities, associated with increased morbidity secondary to implant. This phenomenon is not predictable and its mechanism remains unexplained. The objective of this STREAM study is to generate longitudinal clinical and imaging data on the Silk Vista to further evaluate its efficacy and safety in the treatment of unruptured IA, and in particular, to assess and understand the impact of morphological changes over time associated with this device

DETAILED DESCRIPTION:
Intracranial aneurysms (IA) are abnormal outpouchings of cerebral arteries' walls. IA prevalence ranges between 1.8% and 8% in adults, with an approximately equal male/female distribution and a mean age of 50 years at first detection. They predominantly occur in arteries found in the Circle of Willis and the middle cerebral artery bifurcation (85%). The primary concern after discovery of an unruptured IA (UIA) is the risk of rupture leading to subarachnoid hemorrhage (SAH) and potentially death. The aneurysmal SAH has been associated with up to 50% mortality, whereas approximately 30% of survivors are left with severe neurological and/or neurocognitive deficits, resulting in a significant public health burden. Given the evidence that when an IA is treated before rupture, survival rates improve dramatically, identification of aneurysms, specifically those at risk of rupture, and availability of effective treatment strategies, are essential for improving the clinical outcomes of these patients. The IA treatment management includes surgery (neurosurgical clipping has been the gold standard) or endovascular methods. However, over the past decade, the endovascular options to manage IA, ruptured or not, have rapidly evolved, making the treatment of IA less invasive and increasingly more successful. In endovascular technique, a parent artery reconstruction is realized with a flow-diverter stent. Following their specific characteristics, flow diverters (FD) were initially designed to treat giant and large. When comparing FD to the other endovascular techniques (coiling or stenting), FD have been shown to have a higher rate of occlusion for large aneurysms. However, during follow-up, up to 15% of FD present a stenosis that may affect their extremities (known as " fishmouth " stenosis) or their mid-segment (" stent collapse "). The deformities are associated with increased morbidity secondary to implant. This phenomena is not predictable and its mechanism remains unexplained. The DFT (drawn-filled tubing with platinum) technology used for braiding the latest generation of FD stents, including the SILK VISTA stent, may potentially contribute to this phenomenon. Data from an independent and comprehensive evaluation are needed to confirm safety and efficacy in this context. The Silk Vista SDF (BALT, Montmorency, France) is intended for the treatment of IA. The objective of this STREAM study is to generate longitudinal clinical and imaging data on the Silk Vista to further evaluate its efficacy and safety in the treatment of UIA, and in particular to assess and understand the impact of morphological changes over time associated with this device.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years old,
* Patient has at least one unruptured intracranial aneurysm intended to be treated with Silk Vista
* Has an untreated or recanalized, unruptured or previously ruptured aneurysm whose rupture occurred >30 days prior to the index procedure
* Able and willing to comply with study procedures including returning to the study site for imaging exams
* Able and willing to give oral informed consent

Exclusion Criteria:

* Any criteria for non- or contraindication to endovascular treatment and/or flow-diverting stent placement (e.g., suspected mycotic aneurysm, including those caused by a left atrial myxoma, systemic bacterial infection, contraindication to antiplatelet drugs (aspirin, clopidogrel/Plavix, ticagrelor, and heparin), local or general anesthesia, allergy to the contrast agent required for treatment by the diversion technique, known severe allergy or hypersensitivity to nickel, titanium, tungsten, or platinum; cost of treatment for an intracranial aneurysm within the last 6 months; and for women, pregnant, or currently breastfeeding)
* Has a true bifurcation aneurysm, defined as an aneurysm (saccular or non-saccular) located at a point of vessel bifurcation
* Has vessel characteristics, such as severe tortuosity, stenosis, or morphology that would preclude safe endovascular access to the target aneurysm necessary for treatment with the study device.
* Presence of intracranial atherosclerotic disease.
* Received previous treatment of the target aneurysm or parent artery where it would interfere with the placement or proper apposition of the device
* Subarachnoid hemorrhage unrelated to a ruptured target aneurysm which occurred within 30 days prior to enrollment
* Intracranial parenchymal hemorrhage occurred within 30 days prior to enrollment
* Major surgery (including previous intracranial implant) occurred within previous 30 days or is planned in the next 6 months after enrollment date
* Has more than one known IA that is anticipated to require treatment within 6 months of the index procedure
* Chronic anticoagulation therapy is ongoing or known coagulopathy exists
* Patient has a serious or life-threatening comorbidity that could confound study results
* Presence of intracranial mass (tumor, except meningioma, abscess, or other infection), non-treated arteriovenous malformation (AVM) in the territory of the target aneurysm
* Participation in any other investigational study which may interfere with collection of valid data under this study or may influence study endpoints Unable to complete study follow up (12 months) due to geographical distance
* Unable to understanding study
* Under legal protection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18 and ≤ 80 years old, with at least one unruptured intracranial aneurysm intended to be treated with Silk Vista
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between stent modification with the geometry of the parent artery and the aneurysm and the dimensions of the stent. | Month 12
  Correlation between stent modification (shortening and/or degree and location of stenosis) with the geometry of the parent artery and the aneurysm and the dimensions of the stent (diameter and length).

SECONDARY OUTCOMES:
Complete occlusion rate | Month 12
  Complete occlusion rate of the intracranial aneurysm. Intracranial aneurysm occlusion is measured using three scales :
  * Cekirge-Saatci : 5 levels from Class 1 (Complete occlusion of the aneurysm sac) to class 5 (Stable remodeling with flow modification)
  * O'Kelly-Marotta : including Aneurysm filling (from A-total filling (>95%) to D-no filling (0%)) and Stasis phase (from 1-no stasis (arterial phase clearance, before capillary phase) to 3-significant stasis (persistent contrast at venous phase))
  * Modified Raymond-Roy : from class I (complete obliteration) to class III (residual aneurysm)
Occlusion level | Month 12
  Occlusion level of the treated aneurysm (acceptable (90-100%); without stenosis of the parent artery (>50%). Intracranial aneurysm occlusion is measured using three scales :
  * Cekirge-Saatci : 5 levels from Class 1 (Complete occlusion of the aneurysm sac) to class 5 (Stable remodeling with flow modification)
  * O'Kelly-Marotta : including Aneurysm filling (from A-total filling (>95%) to D-no filling (0%)) and Stasis phase (from 1-no stasis (arterial phase clearance, before capillary phase) to 3-significant stasis (persistent contrast at venous phase))
  * Modified Raymond-Roy : from class I (complete obliteration) to class III (residual aneurysm)
Successful stent deployment | Month 12
  Successful stent deployment at the target site, defined as the absence of implantation of a new device at the target aneurysm, endovascular treatment, additional stenting, or stent stenosis
disabling stroke | Month 1, Month 6
  Absence of disabling stroke or death (assessed by a Clinical Events Committee).
Major stroke | Day 7
  Occurrence of a major stroke within 7 days post-procedure (NIHSS +4 compared to baseline
Minor stroke | Day 7
  Occurrence of a minor stroke within 7 days post-procedure (complete resolution or increase of less than 3 points on the National Institutes of Health Stroke Scale (NIHSS
Neurological events | Month 12
  Any neurological event (regardless of relationship) leading to clinical deterioration, based on the change in the mRS (modified Rankin Scale) score : If the baseline mRS score is between 0 and 2, a deterioration is considered if it changes between 3 and 5; If the baseline mRS score is between 3 and 5, a deterioration is considered if it increases by one point from the baseline score.
Morphological changes | Month 1, Month 6, Mont 12
  Incidence of morphological changes over the stent period (stent stenosis ≥50%).
Parent artery occlusion | Month 12
  Incidence of parent artery occlusion
Intracranial hemorrhage | Month 1, Month 6, Mont 12
  Incidence of intracranial hemorrhage (aneurysm-related)
Adverse events | Month 1, Month 6, Mont 12
  Incidence of adverse events (other)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No